CLINICAL TRIAL: NCT06696404
Title: The Role of Nerve Block-Constructed Precision Anesthesia on Perioperative Organ Protection in Hip Surgery
Brief Title: The Role of Precision Anesthesia Strategy on Perioperative Organ Protection in Hip Surgery [PASPOP]
Acronym: PASPOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Collaborators: Army Medical Center of PLA (Other Government)
Responsible Party: Principal Investigator, Tao Xu, Dr, Shanghai 6th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024-147-（1）
Record Dates: First submitted 2024-11-07; First posted 2024-11-20 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Elderly (People Aged 65 or More); Hip Fracture; Delirium - Postoperative; Organ Protection; Nerve Block
Keywords: nerve block; hip fracture; elderly; postoperative delirium; organ protection
MeSH Terms: conditions — Hip Fractures; Emergence Delirium | interventions — Anesthesia, Spinal

STUDY DESIGN:
Intervention Model Description: 1. Nerve block anesthesia group (NA group): Combined Lumbar Plexus(0.33% ropivacaine 30ml)and Sacral Plexus Block(0.33% ropivacaine 20ml) + sedation or laryngeal mask anesthesia
  2. General anesthesia group (GA group): General anesthesia (Endotracheal intubation) + iliac fascial block(0.33% ropivacaine 30ml)
  3. Spinal anesthesia group (SA group): Spinal anesthesia with ropivacaine 8-20 mg or an equivalent dose of Bupivacaine.
Who Masked: Outcomes Assessor
Masking Description: The statistician is blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- NA group (Experimental): Nerve block anesthesia group(NA) Intervention: combined Lumbar Plexus and Sacral Plexus Block, with sedation or laryngeal mask anesthesia (induction with Propofol 1-3mg/kg, Sufentanil 0.1-0.4ug/kg)
  Interventions: Procedure: Combined Lumbar Plexus and Sacral Plexus Block
- GA group (Active Comparator): General anesthesia was performed as an endotracheal intubation combined with iliac fascial block (0.33 ropivacaine 30 ml)
  Interventions: Procedure: iliac fascial block
- SA group (Active Comparator): Spinal anesthesia was performed as a standard care of spinal anesthetic
  Interventions: Procedure: spinal anesthesia

INTERVENTIONS:
Procedure: Combined Lumbar Plexus and Sacral Plexus Block — This intervention of Combined Lumbar Plexus and Sacral Plexus Block is assigned to Nerve block anesthesia group (NA group): A combined Lumbar Plexus Block (0.33% Ropivacaine 30ml) and Sacral Plexus Block (0.33% Ropivacaine 20ml) administered as a single injection.
  Other Names: Lumbar - Sacral Plexus Block; Lumbosacral Plexus Block; Lumbosacral Plexus Nerve Block; Lumbosacral Regional Nerve Block; Lumbosacral Plexus Regional Block
  Arms: NA group
Procedure: iliac fascial block — iliac fascial block administered as a single injection below the iliac fascial with 0.33% ropivacaine 30ml.
  Other Names: iliac fascial compartment block; Fascia Iliaca Block; Fascia Iliaca Nerve Block; Fascia Iliaca Block Technique
  Arms: GA group
Procedure: spinal anesthesia — Spinal anesthesia was performed as a standard care of spinal anesthetic. The spinal puncture site is at L2-3 or L3-4. After the puncture needle reaches the subarachnoid space, 1% ropivacaine 0.8-2 ml, totaling 8-20mg, is injected. Depending on the center's practice, it may be replaced with an equivalent dose of bupivacaine .
  Other Names: spinal block; intrathecal anesthesia
  Arms: SA group

SUMMARY:
The goal of this clinical trial is to investigate the effect of three anesthetic strategies on organ protection in elderly patients undergoing hip fracture surgery.

The main questions it aims to answer are: 1.Does the nerve block anesthesia group have a protective effect on the incidence of postoperative delirium in elderly patients undergoing hip surgery? 2.Does the nerve block anesthesia group also provide protective effects on other organs for elderly patients undergoing hip surgery? 3.What effects will these anesthetic strategies have on short-term and long-term prognosis of elderly patients undergoing hip surgery?

The investigators will compare it with the spinal anesthesia group and the general anesthesia group to see which has a better protective effect on organs.

Participants will undergo preoperative interviews and will be interviewed twice daily, in the morning and evening, from postoperative day 1 to 7 or until discharge, to assess the occurrence of delirium and cognitive levels, pain intensity, and sleep status.

Interventions:

1. Nerve block anesthesia group (NA group): Combined Lumbar and Sacral Plexus Block + sedation or laryngeal mask anesthesia
2. General anesthesia group (GA group): General anesthesia (Endotracheal intubation) + iliac fascial block
3. Spinal anesthesia group (SA group): Spinal anesthesia without any nerve blockade

DETAILED DESCRIPTION:
Background: Over 10 million hip fractures happen per year globally, which lead to a burden on patients, their families, and healthcare systems.98% hip fracture patients require orthopedic surgery. Hip fracture patients are typically elderly and often have multiple comorbidities, decreased organ function, poor physical tolerance, high anesthesia risks, and slow postoperative recovery. Perioperative blood loss is considerable during hip surgery, and the stress response is significant, often leading to severe postoperative pain, which can result in organ damage and complications. These patients pose challenges to anesthesia management, but at the same time, making the anesthetic care episode a major opportunity to impact outcomes.In clinical practice, general anesthesia and spinal anesthesia are the two most commonly used anesthesia strategies. However, current domestic and international studies believe that there is no difference in outcomes for patients undergoing hip surgery under these two strategies. With the advancement of medical science, nerve blocks, due to precise action on the surgical area and effective suppression of postoperative pain, are increasingly applied in clinical settings. When combined with light general anesthesia, nerve blocks can meet surgical requirements. Nerve blocks can reduce quadriceps spasms, decrease stress responses, help maintain hemodynamic stability, and thus might have potential organ-protective effects. Due to the inconsistent clinical research outcomes regarding nerve blocks, coupled with a lack of high-quality study results, the investigators plan to conduct this study to explore the anesthetic strategy with the most prognostic improvement value for patients undergoing hip surgery. So, it will fill critical evidence gaps to inform policy and practice.

Purpose: The purpose of this study is to explore, in the real world, which anesthesia strategy has more organ-protective effects and accelerates postoperative recovery for patients undergoing hip surgery.

Research Design: A prospective randomized three-arm parallel-group double-center exploratory trial with blinded end point evaluation.

Primary hypothesis is that participantis who receive combined lumbar plexus and sacral plexus block + sedation or laryngeal mask anaesthesia will demonstrate improved recovery after randomisation compared with participants who receive general anaesthesia or spinal anesthesia.

Research population: Elderly patients with acute hip fractures requiring surgical treatment.

Interventions:

Participants randomly assigned to NA or GA or SA group in a 1:1:1 ratio.

1. Nerve block anesthesia group (NA group): Combined Lumbar Plexus and Sacral Plexus Block + sedation or laryngeal mask anesthesia. Participants assigned to the NA group will receive lumbar-sacral plexus block combined with laryngeal mask anesthesia. The lumbar-sacral plexus block (0.33% ropivacaine 30ml+20ml) will be performed under the guidance of an ultrasound or nerve stimulator, and the effectiveness of the block will be assessed 20 minutes after the nerve block. Subsequently, participants will undergo sedation or laryngeal mask anesthesia.
2. General anesthesia group (GA group): General anesthesia + iliac fascial block .Participants assigned to the GA group will receive iliac fascial block combined with endotracheal intubation general anesthesia. The iliac fascial block (0.33% ropivacaine 30ml) will be performed under the guidance of an ultrasound or nerve stimulator, and the effectiveness of the block will be assessed 20 minutes after the nerve block. Subsequently, participants will undergo endotracheal intubation general anesthesia.
3. Spinal anesthesia group (SA group):Spinal anesthesia without any nerve blockade. Participants assigned to the SA group will receive spinal anesthesia with or without sedation. Spinal anesthesia is The spinal puncture site is at L2-3 or L3-4. After the puncture needle reaches the subarachnoid space, 1% ropivacaine 0.8-2 ml, totaling 8-20mg, is injected. Depending on the center's practice, it may be replaced with an equivalent dose of bupivacaine .

Statistical analysis:

This study employed R Studio software version 4.3.3 (R Project for Statistical Computing) for data analysis. The specific methodologies are detailed below:

Analysis Principles Primary analysis set: Intent-to-treat (ITT) analysis Randomization method: Stratified randomization by study center

Data Distribution Assessment Normality of continuous variables was evaluated using the Shapiro-Wilk test Normally distributed data: Presented as mean ± standard deviation (Mean ± SD) Non-normally distributed data: Presented as median (interquartile range, Median [IQR])

Intergroup comparison methods Continuous variables

For normally distributed data:

Intergroup comparisons among three groups were performed using one-way analysis of variance (ANOVA).

When ANOVA showed significant differences (P < 0.05), pairwise comparisons were conducted using Student's t-test with Bonferroni correction.

For non-normally distributed data:

Intergroup comparisons were performed using the Kruskal-Wallis nonparametric test.

When significant differences were detected, pairwise comparisons were conducted using the Mann-Whitney U test.

Median differences were calculated using Hodges-Lehmann estimators with 95% confidence intervals (95% CI).

Categorical variables were presented as frequency (percentage, n (%)), Intergroup comparisons were performed using chi-square test (χ² test) or Fisher's exact test (for small sample sizes).

Statistical Significance Criteria:

All tests were two-sided, Significance threshold: P < 0.05.

Multiple comparison adjustment: When performing multiple pairwise comparisons, the significance level (α) was adjusted to 0.05/number of comparisons (Bonferroni method)

Study end points will be assessed via in-person interview (during hospitalisation), medical record review, telephone interview(after hospital discharge).

This study is designed as a Pilot study to provide data reference for future large-sample studies. The study plans to include 30 patients per group, totaling 90 patients across three groups.

Statistical Analysis: The statistical analysis software used was SAS 9.4. ① For the primary outcome measures, continuous variables were analyzed and expressed using standard deviation mean or interquartile range median, and the distribution type of the data was assessed for normality. Categorical variables were represented by counts and percentages. A modified intention-to-treat (ITT) analysis was employed. Randomization was stratified by hospital. The risk of the primary outcome was compared within each group. Additionally, the primary outcome measures could also be analyzed using a generalized linear model to adjust for potential confounding factors, Risk Ratio (crude, adjusted), and their 95% CI. The model was adjusted for the type of surgery and sensitivity analysis was performed to clarify the impact of data missingness on the robustness of the model. ② For the analysis of secondary outcome measures, depending on the variable situation, different types of variables were analyzed using generalized linear models, generalized estimating equations, Winratio, and COX regression, respectively.

Analysis of Data: All analyses were two-tailed tests, with a statistically significant difference set at P<0.05.

Expected test progress: 30 days

ELIGIBILITY:
Inclusion Criteria:

1. Aged 65 years and older
2. American Society of Anesthesiologists (ASA) physical status 1 to 3
3. Scheduled for unilateral hip surgery

Exclusion Criteria:

1. Have psychiatric disorders or cognitive impairments, or are unable to understand the scale
2. Have a heart failure history (EF < 40) or a history of AMI in 3 months
3. Complex injuries: multiple fractures, chest, abdomen, pelvic and sacral trauma, head trauma, etc.
4. Combined with respiratory failure or hepatic failure (Child-Pugh C) or renal failure (rely on dialysis treatment)
5. Nerve block contraindication: puncture site infection, peripheral neuropathy, regional anesthetic allergy, etc.
6. Contraindications of intraspinal anesthesia: coagulation dysfunction, thrombocytopenia, intraspinal space occupying, infection of puncture site, etc.
7. Relative contraindications of general anesthesia: known difficult airway, malignant hyperthermia, etc.
8. Enrolled in another randomized clinical trial

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-03-12 (Actual); Study Completion 2025-04-05 (Actual)

PRIMARY OUTCOMES:
Incidence of of postoperative delirium | From enrollment to the seventh day after surgery or before discharge
  Incidence of of postoperative delirium within 7 days or before discharge (whichever comes first) is assessed by 3-Minute Diagnostic Interview for Confusion Assessment Method(3D-CAM) scale. Each item in the 3D-CAM instrument directly informs one of the 4 CAM features in the algorithm that leads to determining the presence or absence of delirium.The CAM algorithm is considered positive if the following features are present: Feature 1) Acute onset or fluctuating course and Feature 2) Inattention and either Feature 3) Disorganized thinking or Feature 4) Altered level of consciousness. Negative indicates that the paticipant did not experience delirium at the time of assessment, which is favorable for the paticipant. Positive indicates that the participant is experiencing delirium at the time of assessment.

SECONDARY OUTCOMES:
Postoperative pain score | From enrollment to the third day after surgery
  Postoperative pain score within 3 days after surgery is assessed by visual analogue scale pain score(during resting and movement ).The Visual Analogue Scale (VAS) for pain assessment is commonly used to quantify the severity of pain experienced by participants. The VAS is a simple, continuous scale that is easy to administer and score. A straight line, usually 10 centimeter (cm) in length, is drawn on a piece of paper or presented on a digital device. The endpoints of the line represent the extremes of pain experienced by participants.The left end of the line is anchored with the phrase "No Pain" (0 cm).The right end of the line is anchored with the phrase "Worst Possible Pain" (10 cm).Participants are asked to mark a point on the line that they feel represents their current level of pain.Lower scores( between 0 to 3 ) indicate less severe pain, while higher scores (4-10) indicate more severe pain.
Consumption of opioid medications | From the start of surgery to the seventh day after surgery or at discharge
  The consumption of opioid medications is calculated by translating the number of times a patient activates a patient-controlled analgesia (PCA) pump and any additional analgesics prescribed postoperatively into equivalent doses of morphine.This method allows for a standardized assessment of opioid usage across different types of medications and formulations, providing a consistent metric for evaluating pain management strategies and outcomes. Smaller amount of opioid comsuption is good for patients.
Central nervous system complications | From the start of surgery to the thirtieth day after surgery
  Central nervous system complications within 30 days after surgery is confirmed by CT, MRI or other imaging evidence. Central nervous system complications includes stroke and transient cerebral ischemia.Stroke is defined as the sudden onset of acute neurological deficits, confirmed by CT, MRI, or other imaging evidence, and requiring medical intervention such as anticoagulant therapy.Transient Ischemic Attack (TIA) is defined as a new onset of acute neurological dysfunction caused by cerebral ischemia, lasting less than 1 hour, with no evidence of acute infarction on imaging studies of the head. Medical interventions such as medication (e.g., antiplatelet agents, lipid-lowering drugs) and interventional surgery are required.
Cognitive function | From enrollment to the thirtieth day after surgery
  Cognitive function within 30 days after surgery is assessed by Telephone Montreal Cognitive Assessment(T-MoCA) scale.The T-MoCA is a telephone-based adaptation of the widely recognized Montreal Cognitive Assessment (MoCA), designed to provide a rapid and efficient screening tool for cognitive impairment. It plays a pivotal role in cognitive function assessment by offering a convenient and remote method to evaluate multiple cognitive domains, including attention, concentration, executive functions, memory, language, visuospatial skills, abstraction, calculation, and orientation.The T-MoCA is particularly valuable in diverse community samples, where it has demonstrated sufficient psychometric properties to screen for mild cognitive impairment (MCI), especially in situations where in-person clinic visits are not feasible. A T-MoCA scale less than 18 indicates MCI, and is not good for participants.
Cardiovascular system complications | From enrollment to the thirtieth day after surgery
  Cardiovascular system complications within 30 days after surgery is assessed by through a variety of diagnostic measures. Cardiovascular system complications within 30 days after surgery include myocardial injury, angina, myocardial infarction (heart attack), heart failure, new-onset arrhythmias, and sudden cardiac arrest. Cardiovascular complications are assessed through a variety of diagnostic measures, including elevated troponin levels indicating myocardial injury, symptoms of myocardial ischemia or heart failure, newly diagnosed arrhythmias identified through electrocardiograms (ECGs), and additional evidence from imaging studies such as echocardiograms, nuclear scans, MRI, or CT angiography.
Acute kidney injury (AKI) | From enrollment to the thirtieth day after surgery
  Acute kidney injury (AKI) within 30 days after surgery is assessed using the Kidney Disease: Improving Global Outcomes (KDIGO) scoring system.The KIDGO scoring system is a standardized classification system defines AKI based on changes in serum creatinine levels and urine output. According to the KDIGO guidelines, AKI is defined as any of the following criteria within a 48-hour period: an increase in serum creatinine (SCr) of ≥0.3 mg/dL, or an increase to ≥1.5 times the baseline SCr that is known or presumed to have occurred within the prior seven days, or a urine volume of less than 0.5 mL/kg/hr for six hours.
Inflammatory factors | From enrollment to the third day after surgery
  Inflammatory factors within 3 days after surgery assessed by serum test. Inflammatory indicators include IL-6, CRP, TNF-α etc. Higher inflammatory factors may indicate higher inflammatory response, and is not good for participants.
Other related complications | From enrollment to the thirieth day after surgery
  Other related complications and outcomes within 30 days after surgery assessed via chart review by site staff using standardised outcome definitions, including pulmonary infection, pulmonary edema, hypoxemia, respiratory failure, renal failure, gastrointestinal bleeding,stress ulcer, obstruction etc.
Mortality | From enrollment to the thirtieth day after surgery
  Mortality during hospitalization and 30 days after surgery were obtained through follow-up or telephone-interviews.Data on the mortality outcome were obtained through telephone interviews by trial staff who were unaware of the treatment assignments.
Other outcomes | From enrollment to one year after surgery
  Other outcomes were obtained from follow-up for 1 year of discharge: cognitive function, quality of life, mental condition, mortality via telephone interviewsFollow-up for 1 year of discharge: cognitive function, quality of life, mortality via telephone interviews. Cognitive function is assessed by T-MoCA scale, quality of life is assessed by Activity of Daily Living Scale (ADL scale).

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Arm Medical Center of PLA, Chongqing, Chongqing Municipality
  - Shanghai 6th People's hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided
The data sharing policy is currently under development and is expected to be updated by December 2025.

REFERENCES:
- [Background] Guay J, Kopp S. Peripheral nerve blocks for hip fractures in adults. Cochrane Database Syst Rev. 2020 Nov 25;11(11):CD001159. doi: 10.1002/14651858.CD001159.pub3. PMID 33238043
- [Background] Abou-Setta AM, Beaupre LA, Rashiq S, Dryden DM, Hamm MP, Sadowski CA, Menon MR, Majumdar SR, Wilson DM, Karkhaneh M, Mousavi SS, Wong K, Tjosvold L, Jones CA. Comparative effectiveness of pain management interventions for hip fracture: a systematic review. Ann Intern Med. 2011 Aug 16;155(4):234-45. doi: 10.7326/0003-4819-155-4-201108160-00346. PMID 21844549
- [Background] Kim CH, Yang JY, Min CH, Shon HC, Kim JW, Lim EJ. The effect of regional nerve block on perioperative delirium in hip fracture surgery for the elderly: A systematic review and meta-analysis of randomized controlled trials. Orthop Traumatol Surg Res. 2022 Feb;108(1):103151. doi: 10.1016/j.otsr.2021.103151. Epub 2021 Nov 23. PMID 34826609
- [Background] Cai L, Song Y, Wang Z, She W, Luo X, Song Y. The efficacy of fascia iliaca compartment block for pain control after hip arthroplasty: A meta-analysis. Int J Surg. 2019 Jun;66:89-98. doi: 10.1016/j.ijsu.2018.12.012. Epub 2019 Jan 24. PMID 30685517
- [Background] Gao Y, Tan H, Sun R, Zhu J. Fascia iliaca compartment block reduces pain and opioid consumption after total hip arthroplasty: A systematic review and meta-analysis. Int J Surg. 2019 May;65:70-79. doi: 10.1016/j.ijsu.2019.03.014. Epub 2019 Mar 25. PMID 30922995
- [Background] Memtsoudis SG, Cozowicz C, Bekeris J, Bekere D, Liu J, Soffin EM, Mariano ER, Johnson RL, Go G, Hargett MJ, Lee BH, Wendel P, Brouillette M, Kim SJ, Baaklini L, Wetmore DS, Hong G, Goto R, Jivanelli B, Athanassoglou V, Argyra E, Barrington MJ, Borgeat A, De Andres J, El-Boghdadly K, Elkassabany NM, Gautier P, Gerner P, Gonzalez Della Valle A, Goytizolo E, Guo Z, Hogg R, Kehlet H, Kessler P, Kopp S, Lavand'homme P, Macfarlane A, MacLean C, Mantilla C, McIsaac D, McLawhorn A, Neal JM, Parks M, Parvizi J, Peng P, Pichler L, Poeran J, Poultsides L, Schwenk ES, Sites BD, Stundner O, Sun EC, Viscusi E, Votta-Velis EG, Wu CL, YaDeau J, Sharrock NE. Peripheral nerve block anesthesia/analgesia for patients undergoing primary hip and knee arthroplasty: recommendations from the International Consensus on Anesthesia-Related Outcomes after Surgery (ICAROS) group based on a systematic review and meta-analysis of current literature. Reg Anesth Pain Med. 2021 Nov;46(11):971-985. doi: 10.1136/rapm-2021-102750. Epub 2021 Aug 25. PMID 34433647
- [Background] O'Gara BP, Gao L, Marcantonio ER, Subramaniam B. Sleep, Pain, and Cognition: Modifiable Targets for Optimal Perioperative Brain Health. Anesthesiology. 2021 Dec 1;135(6):1132-1152. doi: 10.1097/ALN.0000000000004046. PMID 34731233
- [Background] Yoshimura M, Shiramoto H, Koga M, Yoshimatsu A, Morimoto Y. Comparing the effects of peripheral nerve block and general anesthesia with general anesthesia alone on postoperative delirium and complications in elderly patients: a retrospective cohort study using a nationwide database. Reg Anesth Pain Med. 2022 May 30:rapm-2022-103566. doi: 10.1136/rapm-2022-103566. Online ahead of print. PMID 35636781
- [Background] Li T, Li J, Yuan L, Wu J, Jiang C, Daniels J, Mehta RL, Wang M, Yeung J, Jackson T, Melody T, Jin S, Yao Y, Wu J, Chen J, Smith FG, Lian Q; RAGA Study Investigators. Effect of Regional vs General Anesthesia on Incidence of Postoperative Delirium in Older Patients Undergoing Hip Fracture Surgery: The RAGA Randomized Trial. JAMA. 2022 Jan 4;327(1):50-58. doi: 10.1001/jama.2021.22647. PMID 34928310
- [Background] Neuman MD, Feng R, Carson JL, Gaskins LJ, Dillane D, Sessler DI, Sieber F, Magaziner J, Marcantonio ER, Mehta S, Menio D, Ayad S, Stone T, Papp S, Schwenk ES, Elkassabany N, Marshall M, Jaffe JD, Luke C, Sharma B, Azim S, Hymes RA, Chin KJ, Sheppard R, Perlman B, Sappenfield J, Hauck E, Hoeft MA, Giska M, Ranganath Y, Tedore T, Choi S, Li J, Kwofie MK, Nader A, Sanders RD, Allen BFS, Vlassakov K, Kates S, Fleisher LA, Dattilo J, Tierney A, Stephens-Shields AJ, Ellenberg SS; REGAIN Investigators. Spinal Anesthesia or General Anesthesia for Hip Surgery in Older Adults. N Engl J Med. 2021 Nov 25;385(22):2025-2035. doi: 10.1056/NEJMoa2113514. Epub 2021 Oct 9. PMID 34623788
- [Background] Griffiths R, Babu S, Dixon P, Freeman N, Hurford D, Kelleher E, Moppett I, Ray D, Sahota O, Shields M, White S. Guideline for the management of hip fractures 2020: Guideline by the Association of Anaesthetists. Anaesthesia. 2021 Feb;76(2):225-237. doi: 10.1111/anae.15291. Epub 2020 Dec 2. PMID 33289066
- [Background] Sciard D, Cattano D, Hussain M, Rosenstein A. Perioperative management of proximal hip fractures in the elderly: the surgeon and the anesthesiologist. Minerva Anestesiol. 2011 Jul;77(7):715-22. Epub 2011 Feb 1. PMID 21283071
- [Background] Vaurio LE, Sands LP, Wang Y, Mullen EA, Leung JM. Postoperative delirium: the importance of pain and pain management. Anesth Analg. 2006 Apr;102(4):1267-73. doi: 10.1213/01.ane.0000199156.59226.af. PMID 16551935
- [Background] Lynch EP, Lazor MA, Gellis JE, Orav J, Goldman L, Marcantonio ER. The impact of postoperative pain on the development of postoperative delirium. Anesth Analg. 1998 Apr;86(4):781-5. doi: 10.1097/00000539-199804000-00019. PMID 9539601
- [Background] Shen Y, Liu W, Zhu Z, Liu S, Cao Y, Yan L, Chen L. Application of a preoperative pain management mode based on instant messaging software in elderly hip fracture patients: a randomized controlled trial. BMC Geriatr. 2023 Mar 30;23(1):186. doi: 10.1186/s12877-023-03905-2. PMID 36991402
- [Background] Foss NB, Kristensen BB, Bundgaard M, Bak M, Heiring C, Virkelyst C, Hougaard S, Kehlet H. Fascia iliaca compartment blockade for acute pain control in hip fracture patients: a randomized, placebo-controlled trial. Anesthesiology. 2007 Apr;106(4):773-8. doi: 10.1097/01.anes.0000264764.56544.d2. PMID 17413915
- [Background] Gou RY, Hshieh TT, Marcantonio ER, Cooper Z, Jones RN, Travison TG, Fong TG, Abdeen A, Lange J, Earp B, Schmitt EM, Leslie DL, Inouye SK; SAGES Study Group. One-Year Medicare Costs Associated With Delirium in Older Patients Undergoing Major Elective Surgery. JAMA Surg. 2021 May 1;156(5):430-442. doi: 10.1001/jamasurg.2020.7260. PMID 33625501
- [Background] Memtsoudis SG, Ma Y, Gonzalez Della Valle A, Besculides MC, Gaber LK, Koulouvaris P, Liu SS. Demographics, outcomes, and risk factors for adverse events associated with primary and revision total hip arthroplasties in the United States. Am J Orthop (Belle Mead NJ). 2010 Aug;39(8):E72-7. PMID 20882208
- [Background] Zhang C, Feng J, Wang S, Gao P, Xu L, Zhu J, Jia J, Liu L, Liu G, Wang J, Zhan S, Song C. Incidence of and trends in hip fracture among adults in urban China: A nationwide retrospective cohort study. PLoS Med. 2020 Aug 6;17(8):e1003180. doi: 10.1371/journal.pmed.1003180. eCollection 2020 Aug. PMID 32760065
- [Background] Witlox J, Eurelings LS, de Jonghe JF, Kalisvaart KJ, Eikelenboom P, van Gool WA. Delirium in elderly patients and the risk of postdischarge mortality, institutionalization, and dementia: a meta-analysis. JAMA. 2010 Jul 28;304(4):443-51. doi: 10.1001/jama.2010.1013. PMID 20664045